CLINICAL TRIAL: NCT05456490
Title: A Phase 1, Double-Blind, Active- and Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Liposomal Bupivacaine 13.3 Administered Via a Single Intrathecal Injection to Healthy Volunteers
Brief Title: Phase 1, Dose Escalation Study to Evaluate of Safety, Pharmacokinetics and Pharmacodynamics of Liposomal Bupivacaine 13.3 Administered Via a Single Intrathecal Injection to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-124
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Pharmacodynamics; Pharmacokinetics; Safety; Efficiency
MeSH Terms: interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The decision to proceed to the next cohort will be made following a full review of the safety, PK, sensory, motor, neurological history and assessment questionnaires, comprehensive neurological exam and Adverse Event data from the current completed cohort(s).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each of the cohorts will be masked as to proceed to subsequent next dose escalation cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposomal Bupivacaine 13.3 (Experimental): Cohort 1 subjects will be dosed 2 mL (26.6 mg) of Liposomal Bupivacaine 13.3.
  Cohort 2 subjects randomized to the Liposomal Bupivacaine 13.3 arm will be dosed 3 mL (39.9 mg) of Liposomal Bupivacaine 13.3.
  Cohort 3 subjects randomized to the Liposomal Bupivacaine 13.3 arm will be dosed 4 mL (53.2 mg) of Liposomal Bupivacaine 13.3.
  Interventions: Drug: Liposomal Bupivacaine 13.3
- Bupivacaine IT (Active Comparator): Cohort 1 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg/ 1 mL) of 0.75% bupivacaine.
  Cohort 2 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg/ 1 mL) of 0.75% bupivacaine mixed with 1 mL of preservative free normal saline to create a total volume of solution administered of 3 mL.
  Cohort 3 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg / 1 mL) of 0.75% bupivacaine mixed with 2 mL of preservative free normal saline to create a total volume of solution administered of 4 mL.
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): Cohort 1 subjects randomized to the placebo arm will be dosed 2 mL of preservative free normal saline.
  Cohort 2 subjects randomized to the placebo arm will be dosed 3 mL of preservative free normal saline.
  Cohort 3 subjects randomized to the placebo arm will be dosed 4 mL of preservative free normal saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Liposomal Bupivacaine 13.3 — Injection into the Intrathecal space
  Arms: Liposomal Bupivacaine 13.3
Drug: Bupivacaine — Injection into the Intrathecal space
  Arms: Bupivacaine IT
Other: Placebo — Injection into the Intrathecal space
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Primary Objective: To assess the safety and tolerability of Liposomal Bupivacaine 13.3 administered as a single intrathecal injection in healthy volunteers.

Secondary Objective: To characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of Liposomal Bupivacaine 13.3 administered as a single intrathecal injection in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase-1, single center, randomized, double-blind, active and placebo-controlled study in approximately 54 adult healthy subjects (Cohort 1, Cohort 2, and Cohort 3). Eighteen subjects will be enrolled in each of the 3 cohorts.

Subjects in Cohort 1, Cohort 2, and Cohort 3 will be randomized 1:1:1 with 6 subjects receiving Liposomal Bupivacaine 13.3 intrathecal (IT), 6 subjects receiving bupivacaine IT, and 6 subjects receiving placebo IT in each cohort.

The dose of Liposomal Bupivacaine 13.3 (and volume of injectate across all three treatment arms) will be determined by the cohort. Cohort 1 subjects randomized to the Liposomal Bupivacaine 13.3 arm will be dosed 2 mL (26.6 mg) of Liposomal Bupivacaine 13.3, Cohort 2 subjects randomized to the Liposomal Bupivacaine 13.3 arm will be dosed 3 mL (39.9 mg) of Liposomal Bupivacaine 13.3, and Cohort 3 subjects randomized to the Liposomal Bupivacaine 13.3 arm will be dosed 4 mL (53.2 mg) of Liposomal Bupivacaine 13.3.

The dose of bupivacaine IT administered in all cohorts will be 15 mg. Cohort 1 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg/ 1 mL) of 0.75% bupivacaine. Cohort 2 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg/ 1 mL) of 0.75% bupivacaine mixed with 1 mL of preservative free normal saline to create a total volume of solution administered of 3 mL. Cohort 3 subjects randomized to the bupivacaine arm will be dosed 2 mL (7.5 mg / 1 mL) of 0.75% bupivacaine mixed with 2 mL of preservative free normal saline to create a total volume of solution administered of 4 mL.

Cohort 1 subjects randomized to the placebo arm will be dosed 2 mL of preservative free normal saline. Cohort 2 subjects randomized to the placebo arm will be dosed 3 mL of preservative free normal saline. Cohort 3 subjects randomized to the placebo arm will be dosed 4 mL of preservative free normal saline.

The decision to proceed to the next cohort will be made following a full review of the safety, PK, sensory, motor, neurological history and assessment questionnaires, comprehensive neurological exam and Adverse Event data from the current completed cohort(s).

All subjects will remain in the Early Phase Research Unit (EPRU) for 5 days after drug administration and will be discharged on Day 6. Subjects will be instructed to return to the research facility for a Day 9 follow-up visit. Subjects will also receive a phone call on Day 30 (±3 days) to assess safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages ≥18 and ≤50 years old.
2. American Society of Anesthesiologists physical status 1
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine, NSAIDs, spinal anesthesia).
2. Impaired renal or hepatic function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase level >1.5 times the upper limit of normal [ULN], or serum alanine aminotransferase level >1.5 times the ULN).
3. Subjects at an increased risk for bleeding or who have a coagulation disorder (defined as platelet count less than 80,000 × 103/mm3).
4. Subjects with a history of a difficult airway or a potential difficult airway based on exam by an anesthesiologist.
5. Subjects with a history of migraine, cluster, or tension headache (diagnosed by a healthcare provider) at any time over the life-course.
6. Subjects without a formal headache diagnosis, but currently experiencing frequent headaches (of any severity), defined as headache occurring > or = 1 time per week for the last 3 months. Subjects who report hormonal headaches occurring during their monthly menstrual cycle that are not diagnosed by a healthcare provider (e.g., pure menstrual migraine without aura, menstrually-related migraine without aura, pure menstrual migraine with aura, menstrually-related migraine with aura) will be excluded if there is a reported pattern of headaches that occur consistently or most of the time during or before their monthly menstrual period. Note: if a subject reports hormonal headaches that are not diagnosed by a healthcare provider, the subject may be included in the study if the headache episodes are infrequent (e.g., one episode in the past 3 months), at the discretion of the Principal Investigator.
7. Subjects with a history of a lower back condition (e.g., ankylosing spondylitis, scoliosis, dysraphism, prior back surgery) or a history of chronic low back pain.
8. Subjects with BMIs less than 20 kg/m2.
9. Comorbidity impacting current physical function that, in the opinion of the investigator, may confound the post dosing assessments
10. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which may confound the post dosing assessments.
11. Women of childbearing potential must have a documented negative pregnancy test at screening and must be confirmed on the day of drug administration. If postmenopausal, must have a documented follicle stimulating hormone test confirming menopause at screening.
12. Currently pregnant, nursing, or planning to become pregnant during the study.
13. Clinically significant abnormal ECG that in the opinion of the investigator would preclude the subject from participation in the study.
14. Previous participation in a Pacira sponsored study.
15. Use of systemic corticosteroids up to 3 days prior to study drug administration.
16. Initiation of treatment with neuromodulating agents (e.g., gabapentin, pregabalin [Lyrica], duloxetine [Cymbalta] etc.) within 1 month prior to Screening or ongoing concomitant use if use is for pain control. a. Subject will be excluded if on neuromodulating agents for chronic pain management. Note: if a subject is on a neuromodulating agent for a reason other than pain control (e.g., a depressive disorder), he or she must be on a stable dose for at least 1 month prior to Screening to be included in the study
17. Opioid medications and NSAIDs are not permitted up to 3 days prior to study drug administration.
18. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
19. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-versus-time curve (AUC0-last and AUC0- ∞) | 7-8 weeks
  Pharmacokinetic Endpoint
Maximum plasma concentration (Cmax) | 7-8 weeks
  Pharmacokinetic Endpoint
Time of Cmax (Tmax) | 7-8 weeks
  Pharmacokinetic Endpoint
The apparent terminal elimination half-life (t1/2el) | 7-8 weeks
  Pharmacokinetic Endpoint
Apparent clearance (CL/F) | 7-8 weeks
  Pharmacokinetic Endpoint
Apparent volume of distribution (Vd) | 7-8 weeks
  Pharmacokinetic Endpoint

SECONDARY OUTCOMES:
Average time to onset of sensory block and motor block | 7-8 weeks
  Pharmacodynamic Endpoint
Average duration of sensory block and motor block | 7-8 weeks
  Pharmacodynamic Endpoint

OTHER OUTCOMES:
Incidence of treatment-emergent AEs (TEAEs) through Day 9 | 7-8 weeks
  Safety Endpoint
Proportion of subjects who have any of the neurological events. | 7-8 weeks
  Safety Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Zaets, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No